CLINICAL TRIAL: NCT05862597
Title: Post COVID-19 syndrome-the Correlation With Suboptimal Health Status and Its Changes of Pulse Diagnosis and Autonomic Nervous System
Brief Title: Post COVID-19 Syndrome Study With Questionnaires and Instruments Measurements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2023-01-023AC
Record Dates: First submitted 2023-03-20; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Detection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Status: Normal examination in recent six months and not fit inclusion criteria of suboptimal health status.
  Interventions: Diagnostic Test: HRV and Pulse diagnosis
- Post-Covid syndrome: (A) Age between 20-70 years old, male or female. (B) Have a history of Covid-19 infection. (C) It has been 3 months since the day when the rapid screening test was negative. Antigen positive turn to negative (D) At least one symptom that cannot be explained by other diagnoses and lasts for at least 2 months after being infected with Covid-19.
  Interventions: Diagnostic Test: HRV and Pulse diagnosis

INTERVENTIONS:
Diagnostic Test: HRV and Pulse diagnosis — Palpation of the 6 pulse positions (right cun, right guan, right chi, left cun, left guan, left chi) measured by the pulse diagnostic instrument.

SUMMARY:
COVID-19 has caused various long-term symptoms affecting different bodily functions. A study shows that traditional Chinese medicine can balance the human body disorder after a virus infection and restore health. The study proposes using pulse diagnosis and cardiac rhythm instruments for disease diagnosis and analysis, decomposing time domain pulse wave signals into different frequency ranges and calculating the "spectral energy ratio" and EP to quantify the patient's pathological pulse. The method has been applied to pulse wave analysis of people with suboptimal health status, and its effectiveness has been preliminarily confirmed. The study aims to find the relationship between these parameters and clinical subjective scale scores, to establish an objective data bridge for Chinese and Western medicine diagnosis. In the future, the analysis method will include more subject data to verify the completeness of the method and establish a feasible prediction model.

DETAILED DESCRIPTION:
The coronavirus pneumonia (COVID-19) epidemic has a major global impact since 2019. So far, due to the continuous emergence of mutated strains of the virus, in addition to different clinical symptoms, the causes of disease and prognosis of infected patients are also different. With the rapid increase in the number of confirmed cases in Taiwan, we can see that there are many sequelae caused by the COVID-19. Although most of the infected patients can fully recover, some people have various medium and long-term symptoms, which are called "Long COVID or Post COVID". In addition to causing lung tissue damage and inflammation, the COVID-19 also affects the digestive system, causing patients to experience symptoms such as diarrhea, vomiting, and loss of appetite; damages the nervous system, causing insomnia, poor memory, and loss of taste and smell; affects the kidneys function and cause edema, etc.; or even reduce the number of sperm cells in men, thereby affecting reproductive function. It can be seen clinically that some symptoms will last for a long time or appear repeatedly. These symptoms may be present at the time of initial infection, may appear after recovery, or recur over time, affecting the patient's daily life. From our study, it reveals that through the conditioning diagnosis and treatment of traditional Chinese medicine, the human body disorder after virus infection can be balanced as soon as possible and the health can be restored.

This research proposes to use pulse diagnosis instrument and cardiac rhythm instrument for disease diagnosis and analysis, decompose time domain pulse wave signal into time domain signals of different frequency ranges, and extract 0-10Hz low frequency wave, 0-50Hz global wave, 13-50 Hz high-frequency waveform calculates the "spectral energy ratio (SER)" and EP to quantify the patient's pathological pulse. Try to find the relationship between this set of parameters and clinical subjective scale scores. The analysis method proposed in this study has been applied to the pulse wave analysis of people with suboptimal health status (SHS), and its effectiveness has been preliminarily confirmed. Corresponding relationship with heart rate variability (heart rate variability, HRV) high and low frequency parameters, to further link the activation status of sympathetic nerve and parasympathetic nerve, and establish an objective data bridge for Chinese and Western medicine diagnosis. In the future, more subject data will be included to verify the completeness of the analysis method and establish a feasible prediction model.

ELIGIBILITY:
Inclusion Criteria:

Adults the age between 20-70 years old with a history of Covid-19 infection,have been an interval of 3 months from the day when the rapid screening test was negative and have some unexplained symptom after being infected with Covid-19 and last for at least 2 months.

Exclusion Criteria:

1. Patient characteristics: have been diagnosed with Covid-19 within seven days, positive in the rapid test,pregnant women or take drugs that could easily affect the heart rate, such as β-Blocker, etc., or installed a pacemaker.
2. Disease characteristics: Subjects who have been diagnosis of mental illness by doctors,or diseases such as cancer that fall under the scope of major diseases covered by the national health insurance .

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have at least one symptom that cannot be explained by other diagnoses and lasts for at least 2 months after being infected with Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-02-14 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
"Skylark" Pulse Analysis System | 6 sceond
  Palpation of the 6 pulse positions (right cun, right guan, right chi, left cun, left guan, left chi) measured by the pulse diagnostic instrument are read into the processing program, and then the time domain signal of each pulse position is analyzed in sequence .

SECONDARY OUTCOMES:
Post-Acute Covid-19 Syndrome questionnaires | 1 day
  suboptimal health status questionnaire-25, SHSQ-25;Body. Constitution Questionaire,BCQ;Post-COVID-19 Chinese Medicine Constitution and Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ying KUNG, doctor, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Center for Traditional Medicine, Taipei Veterans General Hospital, Taipei County, Taiwan